CLINICAL TRIAL: NCT03159949
Title: Exercise Sprint Snacks: The Effects of Prolonged Rest, Reduced Exertion High-intensity Interval Training (PR-REHIIT) Compared to Standard Reduced Exertion High-intensity Interval Training (REHIIT).
Brief Title: Sprint Snacks: The Effects of Prolonged Rest on Reduced Exertion Interval Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H17-00641
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Cardiorespiratory Fitness
Keywords: VO2max, maximal oxygen uptake

STUDY DESIGN:
Masking Description: Participants will know what exercise group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR- REHIIT (Experimental): PR-REHIIT participants ("Sprint Snacks") will participate in 3 separate training session per day on 3 days per week (i.e., 9 sessions per week). Each session lasts 3 minutes and 20 seconds and consists of a two-minute warm-up, a 20-second "all-out" sprint, and a one-minute cool-down. There will be 1-4 hours of rest in between training sessions where participants are free to leave the lab and go about their normal day.
  Interventions: Other: PR-REHIIT
- REHIIT (Experimental): REHIIT participants will come into the lab one time per training days (3 training days per week), each session lasting 10 minutes. Training sessions involve a two-minute warm-up, 3 X 20-second sprints with three minutes rest in between, and a one-minute cool-down.
  Interventions: Other: REHIIT

INTERVENTIONS:
Other: REHIIT — REHIIT participants will come into the lab one time per training days (3 training days per week), each session lasting 10 minutes. Training sessions involve a two-minute warm-up, 3 X 20-second cycling sprints on an exercise bike with three minutes rest in between, and a one-minute cool-down.
  Arms: REHIIT
Other: PR-REHIIT — PR-REHIIT participants will come into the lab on 3 separate occasions on the training days, which occur 3 days per week (i.e., 9 sessions per week). Each session lasts 3 minutes and 20 seconds and consists of a two-minute warm-up, a 20-second "all-out" sprint on a cycle ergometer, and a one-minute cool-down. There will be 1-4 hours of rest in between training sessions where participants are free to leave the lab and go about their normal day.
  Arms: PR- REHIIT

SUMMARY:
An adapted sprint interval training protocol involving 2-3 repeated 20-second sprints separated by 2-3 minutes rest (termed reduced exertion high- intensity interval training (REHIIT)) has been developed and has been shown to promote fitness benefits. This data shows how little exercise one may need to improve cardiorespiratory fitness, provided they are willing to work very hard. However, it is unknown whether the benefits of REHIIT are because of the "all-out" nature of the sprint efforts themselves or the pattern of completing sprints with relatively short (i.e., minutes) rest periods within a workout session.

We are inquiring whether performing the same number and style of sprints with prolonged rest (i.e., 1-4 hours of rest in between sprints) is equally effective for improving aerobic fitness when compared to more traditional sprint interval training with 2-3 minutes of rest between sprints. Such information may make the effectiveness of sprint training more accessible and approachable for individuals unwilling or unable to plan a purposeful REHIIT exercise session into their day. If the rest interval could be prolonged then it may be possible to perform a few sprints as "exercise snacks" throughout the day without the need for a structured interval training session.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive (2 or less bouts of purposeful exercise per week)

Exclusion Criteria:

* If your doctor has informed you that you have a heart condition and should only do physical activity recommended by a doctor.
* If you feel pain in your chest when you perform any physical activity.
* If in the past the month you have had chest pain when you were not doing any physical activity.
* If you lose your balance or consciousness because of dizziness.
* If you have bone or joint problem (for example, back, knee, or hip) that could be made worse by a change in your physical activity.
* If you are currently pregnant or planning on becoming pregnant in the next 6 weeks.
* You have previously had a heart attack or stroke
* You are currently engaging in high-intensity interval training.
* You are currently physically active (engaging in 3 or more bouts of purposeful exercise per week; a "bout" is defined as structured, planned exercise lasting at least 30 minutes)
* You have severe chest pain or blood pressure over 240/140 during baseline testing.
* You have exercise induced asthma or a history of syncope.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Change in VO2max | Before and after the 6 week intervention
  Maximal oxygen uptake assessed using a ramp increase protocol on a cycle ergometer.

SECONDARY OUTCOMES:
Change in 10 km Time Trial Performance | Before and after the 6 week intervention
  Time to complete a simulated 10 km Time Trial on a Cycle ergometer

OTHER OUTCOMES:
Exercise Enjoyment Scale | 6 weeks
  This outcome will measure the enjoyment from either PR-REHIIT or REHIIT exercise intervention
Intention Questionnaire | 6 weeks
  This outcome will measure the likelihood of an individual incorporating either PR-REHIIT or REHIIT into their exercise routine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Individual data will be shown in all manuscript figures